CLINICAL TRIAL: NCT05753553
Title: Incidence and Echocardiographic Predictors of HFpEF in High-Risk Population Afferent to Italian Echo-labs Network
Acronym: rEPORt
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Francesco Bandera, Principal Investigator, IRCCS Policlinico S. Donato
Other Study IDs: 108/int/2019
Record Dates: First submitted 2023-02-17; First posted 2023-03-03 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Heart Failure; Heart Failure With Preserved Ejection Fraction
Keywords: Echocardiographic Predictors; Heart Failure with Preserved Ejection Fraction
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Heart Failure with preserved Ejection Fraction (HFpEF): After signing informed consent, clinical and echocardiographic data will be collected. Thereafter, they will be followed up for major clinical events (cardiovascular death, HF requiring hospitalization, myocardial infarction, and atrial fibrillation) for a period of 12 months.

SUMMARY:
The evolving definitions of HF, the increasing attention of the medical community, and the aging of the population are some of the factors contributing to a still debated incidence and prevalence of HFpEF across the general and specific populations. Despite the current decline in new HF cases, HFpEF shows stable incidence according to epidemiological studies. Cardiovascular risk factors, such as a long history of hypertension, diabetes, obesity, and others seem to be associated with a higher HFpEFincidence. Nevertheless, the potential echocardiographic predictors of HFpEF have not been defined yet.

Hypothesis In a population at high risk for HFpEF, collected using a multicenter echo-lab network, the real incidence of HFpEF cases and echocardiographic predictors can be identified.

Aim 1: to define the incidence of HFpEF in a high-risk cohort of patients afferent to the Italian echo-lab network.

Aim 2: to explore the standard (2D and Doppler data) and advanced (LV and LA strain) echocardiographic parameters associated with and potential predictors of HFpEF.

Methods This is a multicenter, prospective, observational study involving an Italian echo labs network. According to inclusion and exclusion criteria, patients will be enrolled during standard echocardiographic evaluation. After signing informed consent, clinical and echocardiographic data will be collected. Thereafter, they will be followed up for major clinical events (cardiovascular death, HF requiring hospitalization, myocardial infarct, and atrial fibrillation) for a period of 12 months

ELIGIBILITY:
Inclusion Criteria:

* Age >65 years
* Echocardiographic LV EF >50%
* Diastolic dysfunction at echocardiography of at least grade 1
* LV hypertrophy defined as: linear LV mass >115 in men, >95 g/m2 in women
* Left atrium (LA) enlargement defined as LA volume > 34 mL/ m2

Exclusion Criteria:

* Severe chronic renal failure (GFR <15)
* Severe chronic obstructive pulmonary disease (COPD) (FEV1 <1)
* More than moderate valve disease
* Previous cardiac surgery
* Previous LV EF <40%

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: the population at high risk for Heart Failure with preserved Ejection Fraction, wth the following characteristics:
  * Age >65 years
  * LV EF >50%
  * Diastolic dysfunction at echocardiography of at least grade 1
  * LV hypertrophy defined as linear LV mass >115 in men, >95 g/m2 in women
  * Left atrium (LA) enlargement defined as LA volume > 34 mL/ m2
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-03-02 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
incidence of HFpEF | after 12 months from baseline
  to define the incidence of HFpEF in a high-risk cohort of patients afferent to Italian echo-lab network

SECONDARY OUTCOMES:
predictors of HFpEF | baseline
  to explore the standard (2D and Doppler data) and advanced (LV and LA strain) echocardiographic parameters associated with and potentially predictors of HFpEF.
predictors of HFpEF | after 12 months
  to explore the standard (2D and Doppler data) and advanced (LV and LA strain) echocardiographic parameters associated with and potentially predictors of HFpEF.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Bandera, MD, PhD, Principal Investigator — university cardiology department, IRCCS Policlinico San Donato
Locations (6):
- Italy (6):
  - Azienda Ospedaliero-Universitaria di Bari, Bari
  - IRCCS Policlinico San Donato, Milan
  - Azienda Ospedaliero-Universitaria di Modena, Modena
  - AUSL Romagna, Ravenna
  - Università degli Studi di Siena, Siena
  - Università degli studi di Verona, Verona

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dunlay SM, Roger VL, Redfield MM. Epidemiology of heart failure with preserved ejection fraction. Nat Rev Cardiol. 2017 Oct;14(10):591-602. doi: 10.1038/nrcardio.2017.65. Epub 2017 May 11. PMID 28492288
- [Background] Gerber Y, Weston SA, Redfield MM, Chamberlain AM, Manemann SM, Jiang R, Killian JM, Roger VL. A contemporary appraisal of the heart failure epidemic in Olmsted County, Minnesota, 2000 to 2010. JAMA Intern Med. 2015 Jun;175(6):996-1004. doi: 10.1001/jamainternmed.2015.0924. PMID 25895156